CLINICAL TRIAL: NCT04100291
Title: The Effect of Faecal Microbiota Transplantation in the Treatment of Chronic Pouchitis: A Multicentre, Placebo-controlled, Randomized, Double Blinded Trial
Brief Title: Faecal Microbiota Transplantation in the Treatment of Chronic Pouchitis
Acronym: MicroPouch
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 inclusion difficulties
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MicroPouch
Record Dates: First submitted 2019-09-12; First posted 2019-09-24 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pouchitis; Inflammatory Bowel Diseases; Ulcerative Colitis
Keywords: FMT; Microbiota
MeSH Terms: conditions — Pouchitis; Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Active Comparator): Faecal microbiota transplantation
  Interventions: Other: Faecal microbiota transplantation
- Placebo (Placebo Comparator): Placebo mixture
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Faecal microbiota transplantation — FMT by daily enema with donor faeces
  Arms: FMT
Other: Placebo — Placebo by daily enema with placebo mixture
  Arms: Placebo

SUMMARY:
Patients with the chronic bowel disease pouchitis is disabled by bloody diarrhoea and abdominal pain often followed by fever. Pouchitis is an inflammation in a pouch, a reservoir formed by the small intestine in the management of the chronic inflammatory bowel disease, ulcerative colitis. Chronic pouchitis is a rare disease with a prevalence in Denmark of <1.8 per 10,000 people, mostly younger people (<50 years). The standard treatment for pouchitis is intensive broad-spectrum antibiotics for a longer period. However, the treatment often fails after repeated treatments. Recent studies show that patients with pouchitis have an altered composition of the gut flora, called microbiota, compared to healthy individuals. As shown by several studies, faecal microbiota transplantation (FMT) with administration of faeces from healthy donors can alter the microbiota. Treatment with faecal microbiota transplantation is today known to be the ultimate treatment for antibiotic resistant recurrent bowel infection with the bacteria Clostridium difficile. It is however still uncertain if faecal microbiota transplantation can be used to the treatment of chronic pouchitis.

The study primary aims to investigate if transplantation of faeces from healthy donors administrated as enemas to patients with chronic pouchitis is superior to placebo for the treatment of pouchitis.

The project is designed as a multi-center, double-blinded, randomized, placebo-controlled treatment study. A positive result from the project will result in an improved treatment to pouchitis patients. Moreover, repeated long-lasting broad-spectrum treatments with antibiotic, which carry a high risk of antibiotic resistance in the society, will be avoided.

DETAILED DESCRIPTION:
Hypothesis:

Gut dysbiosis plays a significant causal role in chronic pouchitis. Modulating the gut microbiota using FMT has a clinical effect by inducing clinical remission in patients with chronic pouchitis.

Objective of the study:

The aim of the MicroPouch-trial is to investigate if transplantation (FMT) of faeces from healthy donors to patients with chronic pouchitis is clinical significant to placebo for the treatment of pouchitis.

Study design:

The project is designed as a multi-center, double-blinded, randomized, placebo-controlled treatment study.

Methods:

Faecal microbiota transplantation is performed with faeces from healthy donors. Potential donors are recruited from the Danish Blood Bank. They are screened for a various of infectious diseases by serum analysis (haematology, inflammation, liver and kidney function, HIV, Hepatitis, Cytomegalovirus, Epstein Barr virus and HbA1c) and faeces analysis (calprotectin, Clostridium difficile (PCR), enteric pathogenic bacteria and antibiotic-resistant bacteria, parasites, cysts, and viruses). Furthermore, the potential donors will complete an extensive questionnaire regarding general health, risk factors and medical history, before they can be included as faecal donors in the project. The screening procedure is based on recommendation from the European FMT Working Group.

The transplantation is performed by enemas, which contain either faeces from the faecal donors or placebo.

Initial before the treatment with either donor faeces or placebo, the patient will be invited for serum analysis (CRP, leukocytes) and faecal analysis (calprotectin, Clostridium difficile, enteric pathogenic bacteria), followed by a pouchoscopy with collection of biopsies. Materials from serum- and faecal analysis and biopsies will be stored for later analysis purpose. The patient will further complete questionnaires concerning symptoms and quality of life. The stage of disease will be evaluated based on the acknowledged questionnaire for pouchitis called Pouchitis Disease Activity Index (PDAI) score.

The treatment begins after all the initial examinations, and the patient will be treated during one month. The treatment consists of daily enema infusion, which either contain faeces from the faecal donors or placebo. During the treatment, the patient will daily record symptoms related to pouchitis (diarrhea, abdominal pain, bleeding per rectum, fever, general discomfort) and possible adverse effects to the treatment.

At the end of treatment, the patient will meet to a follow-up examination including serum analysis (CRP, leukocytes) and faecal analysis (calprotectin), pouchoscopy incl. biopsies, and the questionnaires applied before the treatment. Materials from serum- and faecal analysis and biopsies will be stored for later analysis.

The patient will be followed up with serum- and faecal analysis and pouchoscopy after additional 6 and 12 months to evaluate the long term effect of the transplantation. The consumption of antibiotics during the first year will be recorded. In case of lacking effect of faecal microbiota transplantation, the patient is offered standard antibiotic treatment for pouchitis, and will leave the study.

Faecal samples and biopsies collected in the study will be analyzed for the composition of the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a J-pouch
* PDAI ≥ 7
* Established diagnosis of chronic pouchitis (≥3 times of pouchitis within the last year, symptoms more than 4 weeks despite antibiotic treatment)
* Antibiotic treatment for pouchitis (ciprofloxacin and/or metronidazole) within the last year
* Not pregnant or breastfeeding

Exclusion Criteria:

* Immunosuppression
* Pregnancy
* Evidence of intestinal pathogen bacteria in the stool at inclusion visit
* Any severe or newly diagnosed concomitant cardiovascular, hepatic, intestinal, renal, endocrine, pulmonary, dental disease with inflammation or psychiatric disorder, which, in the opinion of the investigator, might have an influence on the patient's compliance or the interpretation of the results
* Probiotic intake within the last 2 weeks prior to study intervention
* Participation in another clinical trial within the previous 30 days before baseline
* Serious food allergies with earlier anaphylactic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving clinical remission assessed by PDAI | 4 weeks
  Clinical remission is defined as PDAI<7

SECONDARY OUTCOMES:
Number of patients achieving clinical response assessed by PDAI | 4 weeks
  Clinical response is defined as reduction of PDAI score >2
Number of patients experience improvement in quality of life assessed by the patient-reported questionnaire SIBDQ | 4 weeks
Number of patients relapsing | 12 months
  Relapse is defined as need for antibiotic treatment for pouchitis
Number of patients with treatment-related adverse events in the FMT group compared to the placebo group | 12 months
Increase of the faecal microbiota biodiversity assessed by alpha-diversity | 12 months
Engraftment of the donor microbiota in the patients assessed by beta-diversity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, Study Chair — Aalborg University Hospital
Locations (2):
- Denmark (2):
  - Department of Gastrointestinal Surgery, Aalborg University Hospital, Aalborg
  - Department of Medical Gastroenterology, Copenhagen University Hospital Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Derived] Kousgaard SJ, Cold F, Halkjaer SI, Petersen AM, Kjeldsen J, Hansen JM, Dall SM, Albertsen M, Nielsen HL, Kirk KF, Duch K, Sonderkaer M, Thorlacius-Ussing O. The Effect of Non-pooled Multidonor Faecal Microbiota Transplantation for Inducing Clinical Remission in Patients with Chronic Pouchitis: Results from a Multicentre, Randomised, Double-blinded, Placebo-controlled Trial [MicroPouch]. J Crohns Colitis. 2024 Nov 4;18(11):1753-1766. doi: 10.1093/ecco-jcc/jjae066. PMID 38708959